CLINICAL TRIAL: NCT01494233
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Determine the Safety and Efficacy of Orally Administered LX1033 in Subjects With Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Brief Title: A Multi-Center Trial to Determine the Safety and Efficacy of LX1033 in Subjects With Diarrhea-Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX1033.1-201-IBS; LX1033.201 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose (Experimental): 500 mg LX1033 two times daily
  Interventions: Drug: 250 mg LX1033 tablets
- Mid dose (Experimental): 500 mg LX1033 three times daily
  Interventions: Drug: 250 mg LX1033 tablets
- High dose (Experimental): 1000 mg LX1033 two times daily
  Interventions: Drug: 250 mg LX1033 tablets
- Placebo (Placebo Comparator): Matching placebo dosing
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: 250 mg LX1033 tablets — 250 mg LX1033 tablets administered orally
  Arms: High dose; Low dose; Mid dose
Drug: Placebo tablet — Matching placebo tablet administered orally
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of LX1033 over a range of dose levels in subjects with diarrhea-predominant Irritable Bowel Syndrome (IBS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18 to 70 years, with diarrhea-predominant IBS (IBS-D) with symptom onset at least 6 months prior to diagnosis
* Two or more days per week with at least one stool with a consistency of Type 6 or 7 (Bristol Stool Form Scale)
* Weekly average of worst abdominal pain in past 24 hours score of greater than or equal to 3.0 using a 0-10 point scale
* Ability to provide written, informed consent

Exclusion Criteria:

* Inability to discontinue any current drug therapy for IBS, with the exception of bulking agents. Subjects will be allowed up to 2 doses of loperamide per week as rescue medication.
* Subjects who score severe abdominal pain (rated 7 or higher) 5 or more days per week
* Concomitant use of opioid analgesic drugs or drugs that affect bowel motility
* Any abnormalities or conditions deemed by the investigator as clinically significant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in stool consistency | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in plasma 5-HIAA levels | 4 weeks
Change from baseline in worst abdominal pain in past 24 hours | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sumen Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (78):
- United States (78):
  - Lexicon Investigational Site, Huntsville, Alabama
  - Lexicon Investigational Site, Tempe, Arizona
  - Lexicon Investigational Site, Tucson, Arizona
  - Lexicon Investigational Site, Little Rock, Arkansas
  - Lexicon Investigational Site, North Little Rock, Arkansas
  - Lexicon Investigational Site, Anaheim, California
  - Lexicon Investigational Site, Encinitas, California
  - Lexicon Investigational Site, Los Angeles, California
  - Lexicon Investigational Site, Oakland, California
  - Lexicon Investigational Site, Orange, California
  - Lexicon Investigational Site, San Diego, California
  - Lexicon Investigational Site, Santa Monica, California
  - Lexicon Investigational Site, Tustin, California
  - Lexicon Investigational Site, Westlake Village, California
  - Lexicon Investigational Site, Littleton, Colorado
  - Lexicon Investigational Site, Wheat Ridge, Colorado
  - Lexicon Investigational Site, Waterbury, Connecticut
  - Lexicon Investigational Site, Boynton Beach, Florida
  - Lexicon Investigational Site, Bradenton, Florida
  - Lexicon Investigational Site, Brooksville, Florida
  - Lexicon Investigational Site, DeLand, Florida
  - Lexicon Investigational Site, Jacksonville, Florida
  - Lexicon Investigational Site, Kissimmee, Florida
  - Lexicon Investigational Site, Lauderdale Lakes, Florida
  - Lexicon Investigational Site, Maitland, Florida
  - Lexicon Investigational Site, Orlando, Florida
  - Lexicon Investigational Site, Port Orange, Florida
  - Lexicon Investigational Site, Tampa, Florida
  - Lexicon Investigational Site, Boise, Idaho
  - Lexicon Investigational Site, Meridian, Idaho
  - Lexicon Investigational Site, Addison, Illinois
  - Lexicon Investigational Site, Chicago, Illinois
  - Lexicon Investigational Site, Rockford, Illinois
  - Lexicon Investigational Site, Wichita, Kansas
  - Lexicon Investigational Site, Bowling Green, Kentucky
  - Lexicon Investigational Site, Lexington, Kentucky
  - Lexicon Investigational Site, Chevy Chase, Maryland
  - Lexicon Investigational Site, Towson, Maryland
  - Lexicon Investigational Site, Brockton, Massachusetts
  - Lexicon Investigational Site, Chesterfield, Michigan
  - Lexicon Investigational Site, Kalamazoo, Michigan
  - Lexicon Investigational Site, Troy, Michigan
  - Lexicon Investigational Site, Jackson, Mississippi
  - Lexicon Investigational Site, Mexico, Missouri
  - Lexicon Investigational Site, Billings, Montana
  - Lexicon Investigational Site, Berlin, New Jersey
  - Lexicon Investigational Site, Albuquerque, New Mexico
  - Lexicon Investigational Site, Great Neck, New York
  - Lexicon Investigational Site, New York, New York
  - Lexicon Investigational Site, Boone, North Carolina
  - Lexicon Investigational Site, Cary, North Carolina
  - Lexicon Investigational Site, Chapel Hill, North Carolina
  - Lexicon Investigational Site, Greensboro, North Carolina
  - Lexicon Investigational Site, High Point, North Carolina
  - Lexicon Investigational Site, Raleigh, North Carolina
  - Lexicon Investigational Site, Winston-Salem, North Carolina
  - Lexicon Investigational Site, Fargo, North Dakota
  - Lexicon Investigational Site, Kettering, Ohio
  - Lexicon Investigational Site, Lima, Ohio
  - Lexicon Investigational Site, Mentor, Ohio
  - Lexicon Investigational Site, Wadsworth, Ohio
  - Lexicon Investigational Site, Norman, Oklahoma
  - Lexicon Investigational Site, Oklahoma City, Oklahoma
  - Lexicon Investigational Site, Eugene, Oregon
  - Lexicon Investigational Site, Mt. Pleasant, South Carolina
  - Lexicon Investigational Site, Chattanooga, Tennessee
  - Lexicon Investigational Site, Austin, Texas
  - Lexicon Investigational Site, El Paso, Texas
  - Lexicon Investigational Site, Lake Jackson, Texas
  - Lexicon Investigational Site, Plano, Texas
  - Lexicon Investigational Site, San Antonio, Texas
  - Lexicon Investigational Site, Clinton, Utah
  - Lexicon Investigational Site, Logan, Utah
  - Lexicon Investigational Site, Ogden, Utah
  - Lexicon Investigational Site, Sandy City, Utah
  - Lexicon Investigational Site, West Jordan, Utah
  - Lexicon Investigational Site, Lynchburg, Virginia
  - Lexicon Investigational Site, Virginia Beach, Virginia

REFERENCES:
- [Derived] Delgado-Herrera L, Lasch K, Zeiher B, Lembo AJ, Drossman DA, Banderas B, Rosa K, Lademacher C, Arbuckle R. Evaluation and performance of a newly developed patient-reported outcome instrument for diarrhea-predominant irritable bowel syndrome in a clinical study population. Therap Adv Gastroenterol. 2017 Sep;10(9):673-687. doi: 10.1177/1756283X17726018. Epub 2017 Aug 24. PMID 28932269